CLINICAL TRIAL: NCT03075267
Title: A Phase I, Randomized, Double-Blind, Parallel-Group, Study to Assess the Pharmacokinetics and Safety of Two Doses of PT010 and a Single Dose of PT003 in Healthy Chinese Adult Subjects Following A Single Administrations and After Chronic Administration for 7 Days
Brief Title: Pharmacokinetics and Safety Study of PT010 and PT003 in Healthy Chinese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT010010
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Results first posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- PT010 (BGF MDI) 320/14.4/9.6 µg (Experimental): PT010 Budesonide, Glycopyrronium and Formoterol Fumurate Metered Dose Inhaler (BGF MDI) 320/14.4/9.6 µg
  Interventions: Drug: PT010 (BGF MDI) 320/14.4/9.6 µg
- PT010 (BGF MDI) 160/14.4/9.6 µg (Experimental): PT010 (BGF MDI) 160/14.4/9.6 µg
  Interventions: Drug: PT010 (BGF MDI) 160/14.4/9.6 µg
- PT003 (GFF MDI) 14.4/9.6 µg (Experimental): PT003 (GFF MDI) 14.4/9.6 µg
  Interventions: Drug: PT003 (GFF MDI) 14.4/9.6 µg

INTERVENTIONS:
Drug: PT010 (BGF MDI) 320/14.4/9.6 µg — A single dose of study drug will be administered on Day 1 and BID doses will be administered Day 2 through Day 7 of the Treatment Period, with a final single administration of study drug occurring on the morning of Day 8.
  Other Names: Budesonide, Glycopyrronium, Formoterol Metered Dose Inhaler
  Arms: PT010 (BGF MDI) 320/14.4/9.6 µg
Drug: PT010 (BGF MDI) 160/14.4/9.6 µg — A single dose of study drug will be administered on Day 1 and BID doses will be administered Day 2 through Day 7 of the Treatment Period, with a final single administration of study drug occurring on the morning of Day 8.
  Other Names: Budesonide, Glycopyrronium, Formoterol Metered Dose Inhaler
  Arms: PT010 (BGF MDI) 160/14.4/9.6 µg
Drug: PT003 (GFF MDI) 14.4/9.6 µg — A single dose of study drug will be administered on Day 1 and BID doses will be administered Day 2 through Day 7 of the Treatment Period, with a final single administration of study drug occurring on the morning of Day 8.
  Other Names: Glycopyrronium and Formoterol Fumurate Metered Dose Inhaler
  Arms: PT003 (GFF MDI) 14.4/9.6 µg

SUMMARY:
A study to assess the pharmacokinetics and safety of two doses of PT010 and a single dose of PT003 in healthy Chinese adult subjects

DETAILED DESCRIPTION:
A Phase I, Randomized, Double-Blind, Parallel Group, Study to Assess the Pharmacokinetics and Safety of Two Doses of PT010 and a Single Dose of PT003 in Healthy Chinese Adult Subjects Following a Single Administration and After Chronic Administration for 7 Days

ELIGIBILITY:
Inclusion Criteria:

* Male and female Chinese subjects 18-45 years of age
* Females of childbearing potential must agree to be abstinent or else use one of the medically acceptable forms of contraception A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception.

A male subject with female partner of child bearing potential must agree to use one additional form of medically acceptable contraception

-Be in good general health as assessed at Screening and have no clinically significant abnormal labs at Screening.

Exclusion Criteria:

* Pregnant or nursing female subjects or subjects who are trying to conceive
* Subjects with clinically significant neurologic, cardiovascular, hepatic, renal, endocrinologic, pulmonary, hematological, psychiatric, or other medical illness that would interfere with participation in this study
* Subjects with a history of ECG abnormalities
* Subjects who have cancer that has not been in complete remission for at least 5 years
* Male subjects with symptomatic prostatic hypertrophy that is clinically significant in the opinion of the Investigator
* Male subjects with a trans-urethral resection of the prostate or full resection of the prostate within 6 months prior to Screening
* Males with bladder neck obstruction or urinary retention that is clinically significant in the opinion of the Investigator
* Subjects with a diagnosis of glaucoma that in the opinion of the Investigator has not been adequately treated
* History of substance-related disorders within 1 year of Screening
* History of smoking or the use of nicotine containing products or electronic cigarettes within 3 months of Screening by self-reporting
* A positive alcohol breathalyzer or urine drug screen for drugs of abuse at the Screening Visit or at the beginning of each inpatient period
* Treatment with any prescription or non-prescription drugs (including vitamins, herbal, and dietary supplements) within 30 days
* Positivity for human immunodeficiency virus (HIV) or Hepatitis B surface antigen (HbsAg) or positive hepatitis C antibody at Screening
* Positive for Syphilis Antibody
* Subjects with any flu-like syndrome or other respiratory infections
* Recently vaccinated with an attenuated live virus

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M. Dorinsky, MD, Study Director — Pearl Therapeutics
Locations (1):
- Research Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Huang Y, Assam PN, Feng C, Su R, Dorinsky P, Gillen M. Ethnic pharmacokinetic comparison of budesonide/glycopyrrolate/formoterol fumarate metered dose inhaler (BGF MDI) between Asian and Western healthy subjects. Pulm Pharmacol Ther. 2020 Oct;64:101976. doi: 10.1016/j.pupt.2020.101976. Epub 2020 Nov 2. PMID 33152467
- [Derived] Chen Q, Hu C, Yu H, Shen K, Assam PN, Gillen M, Liu Y, Dorinsky P. Pharmacokinetics and Tolerability of Budesonide/Glycopyrronium/Formoterol Fumarate Dihydrate and Glycopyrronium/Formoterol Fumarate Dihydrate Metered Dose Inhalers in Healthy Chinese Adults: A Randomized, Double-blind, Parallel-group Study. Clin Ther. 2019 May;41(5):897-909.e1. doi: 10.1016/j.clinthera.2019.03.007. Epub 2019 Apr 11. PMID 30982547
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=PT010010&attachmentIdentifier=655b9508-3a4c-48cb-835e-ad569131ecb6&fileName=PT010010-03_China_PK_CSP_v4.0_Redacted-PDF-A.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=PT010010&attachmentIdentifier=aff556d3-330c-4fa8-af1a-1fd3f266eb35&fileName=PT010010_SAP_v1.0_2017-08-24_Redacted-PDF-A.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single site in China.
Pre-assignment Details: Subjects were randomized in a 1:1:1 ratio to 1 of 3 treatments: BGF MDI 320/14.4/9.6 μg, BGF MDI 160/14.4/9.6 μg, or GFF MDI 14.4/9.6 μg.
Groups:
- PT010 (BGF MDI) 320/14.4/9.6 µg: PT010 Budesonide, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (BGF MDI) 320/14.4/9.6 µg
- PT010 (BGF MDI) 160/14.4/9.6 µg: PT010 Budesonide, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (BGF MDI) 160/14.4/9.6 µg
- PT003 (GFF MDI) 14.4/9.6 µg: PT003 Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI) 14.4/9.6 µg
Period: Overall Study
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Started | 32 | 32 | 32
Completed | 31 | 32 | 32
Not Completed | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population - all subjects who received at least 1 dose of any blinded study drug
Units Other Than Participants: Demographics
Groups:
- Total: Total of all reporting groups
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg | Total
Number analyzed (Participants) | 32 | 32 | 32 | 96
Number analyzed (Demographics) | 32 | 32 | 32 | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.1 (3.8) | 26.9 (5.1) | 24.7 (4.1) | 25.6 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 3 | 16
  Male | 25 | 26 | 29 | 80
Race/Ethnicity, Customized [Number; unit: Participants]
  Chinese subjects | 32 | 32 | 32 | 96
Smoking Status [Count of Participants; unit: Participants]
  Non Smoker | 28 | 29 | 30 | 87
  Former Smoker | 4 | 3 | 2 | 9
Weight [Mean (Standard Deviation); unit: kg] | 59.99 (5.29) | 60.00 (6.13) | 62.75 (5.31) | 60.91 (5.68)
BMI [Median (Standard Deviation); unit: kg/m^2] | 21.5 (1.4) | 21.6 (1.2) | 21.9 (1.1) | 21.7 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) - Budesonide
Description: Maximum plasma concentration (Cmax) of Budesonide Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: PK Population - defined as all subjects in the Safety Population who had sufficient data to reliably calculate at least 1 PK parameter and did not have a major protocol deviation
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg
Number analyzed (Participants) | 32 | 32
pg/mL | 459.308 (67.6) | 224.298 (98.1)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) - Budesonide
Description: Maximum plasma concentration (Cmax) of Budesonide Day 8
Time Frame: Day 8 Pre-dose -60, and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg
Number analyzed (Participants) | 31 | 32
pg/mL | 626.435 (78.1) | 315.425 (80.2)

3. Primary Outcome: Maximum Plasma Concentration (Cmax) - Glycopyrronium
Description: Maximum plasma concentration (Cmax) of Glycopyrronium Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 32 | 31 | 31
pg/mL | 4.884 (92.5) | 5.286 (120.8) | 5.674 (113.4)

4. Primary Outcome: Maximum Plasma Concentration (Cmax) - Glycopyrronium
Description: Maximum plasma concentration (Cmax) of Glycopyrronium Day 8
Time Frame: Day 8 Pre-dose -60, and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 31 | 32 | 32
pg/mL | 11.303 (96.9) | 11.754 (103.0) | 13.124 (82.3)

5. Primary Outcome: Maximum Plasma Concentration (Cmax) - Formoterol
Description: Maximum plasma concentration (Cmax) of Formoterol Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 32 | 32 | 32
pg/mL | 9.651 (55.8) | 9.932 (71.9) | 10.618 (76.6)

6. Primary Outcome: Maximum Plasma Concentration (Cmax) - Formoterol
Description: Maximum plasma concentration (Cmax) of Formoterol Day 8
Time Frame: Day 8 Pre-dose -60, and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 31 | 32 | 32
pg/mL | 16.125 (59.1) | 16.945 (54.5) | 17.710 (57.6)

7. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0-12 Hours (AUC 0-12) - Budesonide
Description: Area under the plasma concentration-time curve from 0-12 hours (AUC 0-12) - Budesonide Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg
Number analyzed (Participants) | 32 | 32
h*pg/mL | 1747.910 (43.5) | 811.812 (58.2)

8. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0-12 Hours (AUC 0-12) - Budesonide
Description: Area under the plasma concentration-time curve from 0-12 hours (AUC 0-12) - Budesonide Day 8
Time Frame: Day 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg
Number analyzed (Participants) | 31 | 32
h*pg/mL | 2509.888 (53.4) | 1249.615 (52.0)

9. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0-12 Hours (AUC 0-12) - Glycopyrronium
Description: Area under the plasma concentration-time curve from 0-12 hours (AUC 0-12) - Glycopyrronium Day 1
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 20 | 19 | 20
h*pg/mL | 29.400 (23.5) | 27.197 (41.3) | 29.002 (42.6)

10. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0-12 Hours (AUC 0-12) - Glycopyrronium
Description: Area under the plasma concentration-time curve from 0-12 hours (AUC 0-12) - Glycopyrronium Day 8
Time Frame: Day 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 29 | 28 | 31
h*pg/mL | 69.487 (64.8) | 77.078 (47.5) | 72.636 (57.2)

11. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0-12 Hours (AUC 0-12) - Formoterol
Description: Area under the plasma concentration-time curve from 0-12 hours (AUC 0-12) - Formoterol Day 1
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 32 | 32 | 28
h*pg/mL | 47.843 (35.0) | 46.492 (39.3) | 53.583 (38.0)

12. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0-12 Hours (AUC 0-12) - Formoterol
Description: Area under the plasma concentration-time curve from 0-12 hours (AUC 0-12) - Formoterol Day 8
Time Frame: Day 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 31 | 32 | 32
h*pg/mL | 81.936 (39.5) | 85.322 (34.0) | 83.499 (37.8)

13. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) - Budesonide
Description: Time to maximum plasma concentration (tmax) - Budesonide Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg
Number analyzed (Participants) | 32 | 32
h | 0.333 [0.10 to 2.00] | 0.333 [0.10 to 2.00]

14. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) - Budesonide
Description: Time to maximum plasma concentration (tmax) - Budesonide Day 8
Time Frame: Day 8 Pre-dose -60, and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg
Number analyzed (Participants) | 31 | 32
h | 0.333 [0.10 to 4.00] | 0.333 [0.03 to 4.00]

15. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) - Glycopyrronium
Description: Time to maximum plasma concentration (tmax) - Glycopyrronium Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 32 | 31 | 31
h | 0.100 [0.03 to 2.00] | 0.100 [0.03 to 4.00] | 0.100 [0.03 to 4.00]

16. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) - Glycopyrronium
Description: Time to maximum plasma concentration (tmax) - Glycopyrronium Day 8
Time Frame: Day 8 Pre-dose -60, and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 31 | 32 | 32
h | 0.333 [0.03 to 4.00] | 0.333 [0.03 to 4.00] | 0.333 [0.03 to 2.00]

17. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) - Formoterol
Description: Time to maximum plasma concentration (tmax) - Formoterol Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 32 | 32 | 32
h | 0.833 [0.10 to 2.00] | 0.100 [0.10 to 2.00] | 0.100 [0.10 to 2.00]

18. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) - Formoterol
Description: Time to maximum plasma concentration (tmax) - Formoterol Day 8
Time Frame: Day 8 Pre-dose -60, and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 31 | 32 | 32
h | 0.100 [0.10 to 2.00] | 0.100 [0.10 to 4.00] | 0.100 [0.10 to 4.00]

19. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to the Time of the Last Measurable Plasma Concentration (AUC 0-t) - Budesonide
Description: Area under the plasma concentration-time curve from 0 to the time of the last measurable plasma concentration (AUC 0-t) - Budesonide Day 1
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg
Number analyzed (Participants) | 32 | 32
h*pg/mL | 1884.912 (43.5) | 830.012 (61.1)

20. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to the Time of the Last Measurable Plasma Concentration (AUC 0-t) - Glycopyrronium
Description: Area under the plasma concentration-time curve from 0 to the time of the last measurable plasma concentration (AUC 0-t) - Glycopyrronium Day 1
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 31 | 30 | 28
h*pg/mL | 17.616 (89.8) | 17.707 (111.2) | 20.287 (103.3)

21. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to the Time of the Last Measurable Plasma Concentration (AUC 0-t) - Formoterol
Description: Area under the plasma concentration-time curve from 0 to the time of the last measurable plasma concentration (AUC 0-t) - Formoterol Day 1
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 32 | 32 | 32
h*pg/mL | 48.326 (41.4) | 47.408 (48.2) | 45.950 (78.1)

22. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 Extrapolated to Infinity (AUC 0-∞) - Budesonide
Description: Area under the plasma concentration-time curve from 0 extrapolated to infinity (AUC 0-∞) - Budesonide Day 1
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg
Number analyzed (Participants) | 32 | 32
h*pg/mL | 1936.211 (42.0) | 876.673 (58.8)

23. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 Extrapolated to Infinity (AUC 0-∞) - Glycopyrronium
Description: Area under the plasma concentration-time curve from 0 extrapolated to infinity (AUC 0-∞) - Glycopyrronium Day 1
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 5 | 1 | 3
h*pg/mL | 35.465 (19.6) | 33.014 (NA) — value assessed on only one patient - no coefficient of variation | 43.537 (18.3)

24. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 Extrapolated to Infinity (AUC 0-∞) - Formoterol
Description: Area under the plasma concentration-time curve from 0 extrapolated to infinity (AUC 0-∞) - Formoterol Day 1
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 21 | 18 | 19
h*pg/mL | 61.617 (37.5) | 73.123 (40.5) | 70.608 (46.0)

25. Primary Outcome: Elimination Half-life (t½) - Budesonide
Description: Elimination half-life (t½) - Budesonide Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg
Number analyzed (Participants) | 32 | 32
h | 4.572 (25.3) | 3.168 (31.9)

26. Primary Outcome: Elimination Half-life (t½) - Glycopyrronium
Description: Elimination half-life (t½) - Glycopyrronium Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 20 | 14 | 15
h | 5.676 (52.5) | 8.539 (161.3) | 6.194 (108.2)

27. Primary Outcome: Elimination Half-life (t½) - Formoterol
Description: Elimination half-life (t½) - Formoterol Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 31 | 32 | 28
h | 5.098 (22.7) | 5.657 (38.1) | 5.628 (34.2)

28. Primary Outcome: Apparent Total Body Clearance (CL/F) - Budesonide
Description: Apparent total body clearance (CL/F) - Budesonide Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg
Number analyzed (Participants) | 32 | 32
L/h | 165.271 (42.0) | 182.508 (58.8)

29. Primary Outcome: Apparent Total Body Clearance (CL/F) - Glycopyrronium
Description: Apparent total body clearance (CL/F) - Glycopyrronium Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 5 | 1 | 3
L/h | 406.038 (19.6) | 436.184 (NA) — value assessed on only one patient - no coefficient of variation | 330.757 (18.3)

30. Primary Outcome: Apparent Total Body Clearance (CL/F) - Formoterol
Description: Apparent total body clearance (CL/F) - Formoterol Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 21 | 18 | 19
L/h | 155.801 (37.5) | 131.286 (40.5) | 135.962 (46.0)

31. Primary Outcome: Apparent Volume of Distribution (Vd/F) - Budesonide
Description: Apparent volume of distribution (Vd/F) - Budesonide - Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg
Number analyzed (Participants) | 32 | 32
L | 1090.237 (43.0) | 834.269 (56.2)

32. Primary Outcome: Apparent Volume of Distribution (Vd/F) - Glycopyrronium
Description: Apparent volume of distribution (Vd/F) - Glycopyrronium - Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 5 | 1 | 3
L | 2172.038 (17.6) | 2123.999 (NA) — value assessed on only one patient - no coefficient of variation | 1864.314 (49.8)

33. Primary Outcome: Apparent Volume of Distribution (Vd/F) - Formoterol
Description: Apparent volume of distribution (Vd/F) - Formoterol - Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 21 | 18 | 19
L | 1125.215 (26.0) | 1000.172 (29.2) | 1035.257 (30.9)

34. Primary Outcome: Terminal Elimination Rate Constant (λz) - Budesonide
Description: Terminal elimination rate constant (λz) - Budesonide - Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg
Number analyzed (Participants) | 32 | 32
1/h | 0.152 (25.3) | 0.219 (31.9)

35. Primary Outcome: Terminal Elimination Rate Constant (λz) - Glycopyrronium
Description: Terminal elimination rate constant (λz) - Glycopyrronium - Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 20 | 14 | 15
1/h | 0.122 (52.5) | 0.081 (161.3) | 0.112 (108.2)

36. Primary Outcome: Terminal Elimination Rate Constant (λz) - Formoterol
Description: Terminal elimination rate constant (λz) - Formoterol - Day 1
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 31 | 32 | 28
1/h | 0.136 (22.7) | 0.123 (38.1) | 0.123 (34.2)

37. Primary Outcome: Accumulation Ratio for Cmax (RAC [Cmax]) - Budesonide
Description: Accumulation ratio for Cmax (RAC [Cmax]) - Budesonide
Time Frame: Day 1 Pre-dose and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose and Day 8 Pre-dose -60, and 2, 6, 20, 40 min, 1, 2, 4, 8, 10, 12 and 24 h post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg
Number analyzed (Participants) | 31 | 32
Ratio | 1.400 (71.4) | 1.406 (62.6)

38. Primary Outcome: Accumulation Ratio for Cmax (RAC [Cmax]) - Glycopyrronium
Description: Accumulation ratio for Cmax (RAC [Cmax]) - Glycopyrronium
Time Frame: as for outcome 37
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 31 | 31 | 31
Ratio | 2.383 (86.4) | 2.319 (90.3) | 2.412 (89.7)

39. Primary Outcome: Accumulation Ratio for Cmax (RAC [Cmax]) - Formoterol
Description: Accumulation ratio for Cmax (RAC [Cmax]) - Formoterol
Time Frame: Day 1 and Day 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 31 | 32 | 32
Ratio | 1.678 (50.1) | 1.706 (42.1) | 1.668 (62.2)

40. Primary Outcome: Accumulation Ratio for AUC 0-12 (RAC [AUC 0-12]) - Budesonide
Description: Accumulation ratio for AUC 0-12 (RAC [AUC 0-12]) - Budesonide
Time Frame: Day 1 and Day 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg
Number analyzed (Participants) | 31 | 32
Ratio | 1.455 (45.9) | 1.539 (37.1)

41. Primary Outcome: Accumulation Ratio for AUC 0-12 (RAC [AUC 0-12]) - Glycopyrronium
Description: Accumulation ratio for AUC 0-12 (RAC [AUC 0-12]) - Glycopyrronium
Time Frame: Day 1 and Day 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 18 | 18 | 19
Ratio | 3.324 (47.5) | 3.030 (43.0) | 3.189 (31.5)

42. Primary Outcome: Accumulation Ratio for AUC 0-12 (RAC [AUC 0-12]) - Formoterol
Description: Accumulation ratio for AUC 0-12 (RAC [AUC 0-12]) - Formoterol
Time Frame: Day 1 and Day 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 31 | 32 | 28
Ratio | 1.718 (28.7) | 1.835 (26.2) | 1.620 (27.5)

43. Secondary Outcome: Physical Exam Findings
Description: Number of subjects with clinically significant changes in post baseline physical exam findings
Time Frame: Visit 4, Day 8
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 32 | 32 | 32
Participants
  Significant Findings | 0 | 0 | 0

44. Secondary Outcome: Laboratory Tests
Description: Number of subjects with clinically significant changes in post baseline laboratory tests
Time Frame: Visit 4, Day 8
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 32 | 32 | 32
Participants
  Potassium | 0 | 1 | 0

45. Secondary Outcome: Electrocardiogram
Description: Number of subjects with clinically significant changes in post baseline electrocardiogram
Time Frame: Visit 4, Day 8
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 32 | 32 | 32
Participants
  Significant electrocardiogram changes | 0 | 0 | 0

46. Secondary Outcome: Serious Adverse Events/Adverse Events
Description: Number of subjects with clinically significant changes in post baseline serious TEAEs (treatment-emergent adverse events) or TEAEs leading to withdrawal
Time Frame: Visit 4, Day 8
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 32 | 32 | 32
Participants
  Serious TEAEs/TEAEs leading to withdrawal | 0 | 0 | 0

47. Secondary Outcome: Vital Signs
Description: Number of subjects with clinically significant changes in post baseline vital signs
Time Frame: Visit 4, Day 8
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
Number analyzed (Participants) | 32 | 32 | 32
Participants
  Bradycardia events | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the first administration of study drug through the Final Telephone Follow-up.
Description: The Safety Population was defined as all subjects who receive at least one dose of any blinded study drug. Serious Adverse Events were collected from the first administration of study drug up to 14 days following the last dose of study drug administration.
Arm/Group | PT010 (BGF MDI) 320/14.4/9.6 µg | PT010 (BGF MDI) 160/14.4/9.6 µg | PT003 (GFF MDI) 14.4/9.6 µg
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 14/32 | 11/32 | 14/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PT010 (BGF MDI) 320/14.4/9.6 µg (N=32) | PT010 (BGF MDI) 160/14.4/9.6 µg (N=32) | PT003 (GFF MDI) 14.4/9.6 µg (N=32)
Blood glucose increased (Investigations) | 4 (4) | 3 (3) | 4 (4)
Blood potassium increased (Investigations) | 2 (2) | 1 (2) | 5 (5)
Blood potassium decreased (Investigations) | 2 (3) | 4 (4) | 1 (1)
Bilirubin conjugated increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Blood uric acid increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood glucose decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (3)
Sensation of foreign body (General disorders) | 1 (1) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study site will have the opportunity to publish the results of the study, provided that the sponsor has had the opportunity to review and comment on the study site's proposed publication prior to its being submitted for publication with the prior advice of legal (intellectual property counsel) and with proper regard to the protection of subjects' identities.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT03075267/SAP_000.pdf
  • Study Protocol (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT03075267/Prot_001.pdf